CLINICAL TRIAL: NCT06618885
Title: A Phase 1b, Randomised, Controlled Age De-escalation, Dose-finding Study to Evaluate the Safety, Reactogenicity and Immunogenicity of Full-length MSP1/GLA-SE (SUM-101) Malaria Vaccine in Healthy Young Children, and Infants in Burkina Faso.
Brief Title: Safety and Immunogenicity of SUM-101 Malaria Vaccine in Children and Infants Living in Burkina Faso
Acronym: SUM-101
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: European Vaccine Initiative (Other)
Collaborators: Groupe de Recherche Action en Sante (Other); Luxembourg Institute of Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EVI-CT-001
Record Dates: First submitted 2024-09-23; First posted 2024-10-01 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Malaria,Falciparum
MeSH Terms: conditions — Malaria, Falciparum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This trial will be conducted in a double-blinded manner. Namely, the participants, site staff, sponsor staff, the study monitor(s) and the trial statistician will be blinded to the treatment allocation. The independent statistician and the pharmacist are not blind throughout the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Children (18 months - 5 years) (Experimental): Children (18 months - 5 years) will not be randomised. The first 3 participants will be enrolled as sentinel participants prior to the 6 follower participants. The nine participants of Group 1 will receive three administrations of the SUM-101 vaccine (25µg MSP1 + 5µg GLA-SE) in an open-label design.
  Interventions: Biological: SUM-101
- Infants (5-17 months) (Experimental): For safety reasons, vaccination of infants will be staggered based on the dosage of MSP1 and the GLA-SE adjuvant used. The following dosages will be evaluated:
  * Group 2: 10µg MSP1 + 2.5µg GLA-SE
  * Group 3: 10µg MSP1 + 5µg GLA-SE
  * Group 4: 25µg MSP1 + 2.5µg GLA-SE
  * Group 5: 25µg MSP1 + 5µg GLA-SE Enrollment and vaccination of infants will start with Groups 2 and 3, and only proceed to Groups 4 and 5 if there are no safety concerns. The first infants enrolled into each group will be sentinels (4 per group). The At least tThree out four sentinels will receive the SUM-101 vaccine dose assigned to their respective groups. The participants enrolled into Groups 2-5 (both sentinels and followers) will be randomised at a ratio of 4:1 into vaccine and control arms. In total, 12 participants per group will receive the SUM-101 vaccine (either 25µg or 10µg of MSP1 and either 5µg or 2.5µg of GLA-SE) and 3 participants will receive the control vaccine (rabies vaccine, Verorab®).
  Interventions: Biological: SUM-101

INTERVENTIONS:
Biological: SUM-101 — Three immunizations every 4 weeks for 3 months (total 3 immunizations)

SUMMARY:
This clinical trial aims to learn about the safety and immunogenicity of the blood-stage malaria vaccine candidate SUM-101 in infants and children, paving the way for its incorporation into a multi-stage malaria vaccine. This will be the first time SUM-101 will be evaluated for safety and immunogenicity in infants and children. The main questions it aims to answer are:

* Are the 3 doses of full-length MSP1/GLA-SE (SUM-101) in young children and infants safe?
* Do the 3 doses of full-length MSP1/GLA-SE (SUM-101) in young children and infants produce any reactogenicity?
* How is the immunogenicity in young children and infants generated by the 3 doses of full-length MSP1/GLA-SE (SUM-101)?
* What is the optimal dose of the full-length MSP1/GLA-SE (SUM-101) in young children and infants? The study will be divided into two arms with 5 groups conducted at a single centre. In total, 69 healthy malaria-pre-exposed infants and children aged 5 months to 5 years will be enrolled in this study.

Participants will be included in one of the following groups:

* Arm 1_Group 1 (open-label design): This will be the first cohort enrolled to assess safety in children (18 months - 5 years) before the vaccination of infants commences. Therefore, all participants in Arm 1 will receive three doses of SUM-101 vaccine (25µg MSP1 + 5µg GLA-SE) on D0, D28 and D56.
* Arm 2_Group 2-5 (randomised, controlled, double-blind design): This will be the second cohort enrolled to assess safety in the target population (infants aged 5-17 months). Infants will be assigned to Groups 2-5 to enable evaluation of two doses of MSP1 (25µg and 10µg) and two doses of GLA-SE (5µg and 2.5µg). The infants in each group will be randomised into A) a vaccine arm (12 participants) and B) a control arm (3 participants). All participants in Groups 2-5 will receive three doses of either SUM-101 vaccine or Verorab® (Rabies vaccine) on D0, D28 and D56.

Participants will visit the clinic for screening and once selected for enrolment. No later than 28 days after selection participants will receive the 1st vaccination (Visit Day 0) and 2nd and 3rd Vaccination on Day 28 and Day 56. On Day 1 to 6 days post each vaccination (Day 1-6, Day 29-34 and Day 57-62) each participant will be visited at home daily by a field worker for assessment and recording of any solicited and unsolicited AEs (Reactogenicity visits).

DETAILED DESCRIPTION:
The study will be divided into two arms conducted at a single centre. In total, 69 volunteers will be enrolled in this Phase Ib study to assess the safety, reactogenicity and immunogenicity of SUM-101 in healthy malaria pre-exposed infants and children aged 5 months to 5 years.

Arm 1_Group 1 (open-label design): This will be the first cohort enrolled to assess safety in children (18 months - 5 years) before the vaccination of infants commences. Therefore, all participants in Group 1 (n=9 with n=3 sentinels) will receive three doses of SUM-101 vaccine (25µg MSP1 + 5µg GLA-SE) on D0, D28 and D56 in an open-label design. Female and male participants will be enrolled.

Arm 2_Group 2-5 (randomised, controlled, double-blind design): This will be the second cohort enrolled to assess safety in the target population (infants aged 5-17 months). Infants will be assigned to Groups 2-5 (15 participants in each group with n=4 sentinels) to enable evaluation of two doses of MSP1 (25µg and 10µg) and two doses of GLA-SE (5µg and 2.5µg). To reduce bias, the vaccination of Groups 2-5 will be conducted in a double-blind manner. The infants in each group will be randomised into A) a vaccine arm (12 participants) and B) a control arm (3 participants). Female and male participants will be enrolled. All participants in Groups 2-5 will receive three doses of either SUM-101 vaccine or Verorab® (Rabies vaccine) on D0, D28 and D56.

Sentinel participants: The first 3 participants enrolled in Group 1 will be sentinels who will be vaccinated in an open label manner. To ensure blinding, the first 4 participants enrolled in Groups 2-5 will be sentinels who will be vaccinated with either SUM-101 or control vaccine. The sentinel participants will be vaccinated in the following order; Arm1_Group 1 sentinels: On the first day, the first participant will be enrolled and vaccinated alone and observed on the day following vaccination. If there are no safety concerns, another two participants will be enrolled and vaccinated in a sequential manner at least 48 hours after the first participant and with a minimum interval between participants of 60 min to allow monitoring of any acute events. The remaining participants will be vaccinated at least 72 hours after the third sentinel participant as long as there are no safety concerns.

Arm2_Groups 2-5 sentinels: On the first day, two participants will be enrolled and vaccinated in a sequential manner with a minimum interval between the participants of 60 min to allow monitoring of any acute events. These two vaccinated participants will then be observed on the day following vaccination. If there are no safety concerns, another two participants will be enrolled and vaccinated in a sequential manner at least 48 hours after the first participant and with a minimum interval between participants of 60 min to allow monitoring of any acute events. The remaining participants will be vaccinated at least 72 hours after the fourth sentinel participant as long as there are no safety concerns.

ELIGIBILITY:
Inclusion Criteria:

* Resident in the study area villages and participant's parent(s)/legal guardian anticipate being available for vaccination and follow-up for following last dose of vaccination.
* Z-score of weight-for-age within ±2SD.

Exclusion Criteria:

* Clinically significant skin disorder (psoriasis, contact dermatitis etc.), immunodeficiency, cardiovascular disease, respiratory disease, endocrine disorder, liver disease, renal disease, gastrointestinal disease, neurological illness, major congenital defects, malnutrition requiring hospital admission and anaemia.
* History of allergic reaction, significant IgE-mediated event, or anaphylaxis to immunisation.
* Clinically significant laboratory abnormality as judged by the study investigator.
* History of blood transfusion.
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate.
* Previous vaccination with experimental malaria vaccines.
* Participation in another research study/clinical trial involving receipt of an investigational medicinal product or planned use during the study period.
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection (no HIV testing); asplenia; recurrent, severe infections and chronic immunosuppressant medication (For corticosteroids, this will mean prednisone, or equivalent, 0.5 mg/kg/day. Inhaled and topical steroids are allowed).
* Any significant disease, disorder or situation which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant´s ability to participate in the trial.

Ages: 5 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 69 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Local and systemic solicited adverse events (AEs) at least possibly related to the SUM-101. | After each vaccination (done on Day0, Day28 and Day56) up to 7 days after.
  Local and systemic solicited adverse events (AEs) at least possibly related to the investigational medicinal product (IMP) SUM-101 will be recorded to evaluate safety and reactogenicity.
Local and systemic unsolicited reactogenicity adverse events (AEs). | Recorder after each vaccination (done on Day0, Day28 and Day56) up to 28 days later.
  Local and systemic unsolicited reactogenicity will be recorded to evaluate the safety and reactogenicity of SUM-101.
Number of participants with treatment-related adverse events as assessed by safety laboratory measures of haematology and biochemistry. | Between baseline (Day 0 before 1st vaccination) to 28 days after each vaccination.
  Changes in laboratory safety parameters as summarised as absolute values of:
  Haematology (RBC count, WBC count with differentials (neutrophil, lymphocyte and eosinophil), Haemoglobin (Hgb), Haematocrit and platelet count.
  Biochemistry-, Serum creatinine, Alanine aminotransferase (ALT), Aspartate Aminotransferase (AST) and Total bilirubin.
Any serious adverse events (SAE) occurring during the whole study duration. | Recorded after signature of informed consent until the participant's last visit (Day 140)
  Any serious adverse events (SAE) occurring after signature of the informed consent until the participant's last visit to evaluate the safety and reactogenicity of SUM-101.

SECONDARY OUTCOMES:
IgG antibody titres against full-length MSP1 | Changes assessed between Day 0 (pre-vaccination) up to Day 140 (last follow up visit).
  IgG antibody titters against the full-length MSP1 will be measured by ELISA.
Identification of the dose of full-length MSP1/GLA-SE (SUM-101) in young children and infants that give the safety profile. | Recorded from after 1st vaccination (Day 0 post-vaccination) until the participant's last visit (Day 140)
  Comparison of local and systemic solicited adverse events (AEs) at least possibly related to the investigational medicinal product (IMP) SUM-101 will be recorded to evaluate safety and reactogenicity across different doses of full-length MSP1 and GLA-SE in infants and young children .
Identification of the dose of full-length MSP1/GLA-SE (SUM-101) in young children and infants that give the strongest immune response. | Recorded from after 1st vaccination (Day 0 post-vaccination) until the participant's last visit (Day 140)
  Comparison of IgG antibody titters against the full-length MSP1 will be measured by ELISA across different doses of full-length MSP1 and GLA-SE in infants and young children.

OTHER OUTCOMES:
Evaluation of antibody-mediated complement fixation activity. | Changes assessed between Day 0 (pre-vaccination) up to Day 140 (last follow up visit).
  In vitro immunological assay to evaluate immune responses by assessing complement fixation.
Evaluation of antibody-dependent respiratory burst (ADRB) activity of vaccine-induced antibodies. | Changes assessed between Day 0 (pre-vaccination) up to Day 140 (last follow up visit).
  In vitro lab immunological assay to evaluate immune responses by assessing antibody-dependent respiratory burst (ADRB) activity measured in the sera or blood of all participants.
Age dependency of IgG and IgM antibody titers against full-length MSP1 in comparison to Tanzanian and German adults who previously received SUM-101 vaccine. | Changes assessed between Day 0 (pre-vaccination) up to Day 140 (last follow up visit).
  IgG antibody titters against the full-length MSP1 will be measured by ELISA.
Evaluation of immune-mediated growth inhibition activity on a panel of genetically diverse P. falciparum lines in vitro. | Changes assessed between Day 0 (pre-vaccination) up to Day 140 (last follow up visit).
  In vitro functional assay to evaluate immune-mediated growth inhibition activity on a panel of Plasmodium falciparum asexual blood stage cell lines measured in the sera or blood of all participants.
Evaluation of the opsonic phagocytosis activity of vaccine induced IgG. | Changes assessed between Day 0 (pre-vaccination) up to Day 140 (last follow up visit).
  In vitro immunological assay to evaluate immune responses by measuring opsonic phagocytosis activity in the sera or blood of all participants.
Evaluation of antibody-dependent cellular cytotoxicity (ADCC-NK cells) activity. | Changes assessed between Day 0 (pre-vaccination) up to Day 140 (last follow up visit).
  In vitro immunological assay to evaluate immune responses by assessing antibody-dependent cellular cytotoxicity (ADCC-NK cells) activity in the sera or blood of all participants.
Evaluation of Cytomegalovirus (CMV) seropositivity. | Changes assessed between Day 0 (pre-vaccination) up to Day 140 (last follow up visit).
  In vitro immunological assay to measure CMV seropositivity in comparison with IgG antibody titters against the full-length MSP1 (measured in outcome 5).
Fine-scale resolution of allele-specific antibody responses against full-length MSP1. | Changes assessed between Day 0 (pre-vaccination) up to Day 140 (last follow up visit).
  PepSeq immunology assay to assess allele-specific antibody responses against SUM-101.

CONTACTS AND LOCATIONS:
Overall Officials: Sodiomon Sirima, MD, Principal Investigator — Groupe de Recherche Action en Sante
Locations (1):
- Groupe de Recherche Action en Santé (GRAS), Ouagadougou, Burkina Faso

IPD SHARING:
Plan to Share IPD: No